CLINICAL TRIAL: NCT02642159
Title: A Randomized, Open-Label, Parallel Group Study to Evaluate the Efficacy and Safety of Alirocumab Versus Usual Care in Patients With Type 2 Diabetes and Mixed Dyslipidemia at High Cardiovascular Risk With Non-HDL-C Not Adequately Controlled With Maximally Tolerated Statin Therapy
Brief Title: Efficacy and Safety of Alirocumab Versus Usual Care on Top of Maximally Tolerated Statin Therapy in Patients With Type 2 Diabetes and Mixed Dyslipidemia (ODYSSEY DM-Dyslipidemia)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14354; 2015-001934-19 (EudraCT Number); U1111-1172-5262 (Other: UTN)
Record Dates: First submitted 2015-12-24; First posted 2015-12-30 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-03

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — alirocumab; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe; Fenofibrate; Niacin; Fatty Acids, Omega-3; Hypoglycemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W (Experimental): Alirocumab 75 mg subcutaneous (SC) injection every 2 weeks (Q2W) added to insulin or other antihyperglycemic drugs, stable maximally tolerated dose of statin therapy without other lipid modifying therapy (LMT) for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when non-high-density lipoprotein cholesterol (non-HDL-C) levels >=100 mg/dL (2.59 mmol/L) at Week 8.
  Interventions: Drug: Alirocumab; Drug: Statins; Drug: Antihyperglycemic Drug
- Usual Care (Active Comparator): Participants on usual care continued on insulin or other antihyperglycemic drugs, stable maximally tolerated dose of statin therapy without additional LMT or with either ezetimibe, fenofibrate, omega-3 fatty acids or nicotinic acid as per Investigator's judgment for 24 weeks.
  Interventions: Drug: Statins; Drug: Ezetimibe; Drug: Fenofibrate; Drug: Nicotinic acid; Drug: Omega-3 fatty acids; Drug: Antihyperglycemic Drug

INTERVENTIONS:
Drug: Alirocumab — Solution for injection, one subcutaneous injection in the abdomen, thigh, or outer area of upper arm with a disposable auto-injector.
  Other Names: SAR236553; REGN727; Praluent
  Arms: Alirocumab 75 mg Q2W/Up to 150 mg Q2W
Drug: Statins — Statins at stable dose without other LMT as clinically indicated.
Drug: Ezetimibe — Pharmaceutical form: tablet Route of administration: oral
  Arms: Usual Care
Drug: Fenofibrate — Pharmaceutical form: tablet Route of administration: oral
  Arms: Usual Care
Drug: Nicotinic acid — Pharmaceutical form: tablet Route of administration: oral
  Arms: Usual Care
Drug: Omega-3 fatty acids — Pharmaceutical form: tablet Route of administration: oral
  Arms: Usual Care
Drug: Antihyperglycemic Drug — Insulin (injectable or inhaled) or other antihyperglycemic drugs as clinically indicated.

SUMMARY:
Primary Objective:

To demonstrate the superiority of alirocumab in comparison with usual care in the reduction of non-high-density lipoprotein cholesterol (non-HDL-C) in participants with type 2 diabetes and mixed dyslipidemia at high cardiovascular risk with non-HDL-C not adequately controlled with maximally tolerated statin therapy.

Secondary Objectives:

* To demonstrate whether alirocumab is superior in comparison with usual care in its effects on other lipid parameters (ie, low-density lipoprotein cholesterol (LDL-C), apolipoprotein B (Apo B), total cholesterol (Total -C), lipoprotein a (Lp[a]), high-density lipoprotein cholesterol (HDL-C), triglycerides (TGs), triglyceride rich lipoproteins (TGRLs), apolipoprotein A-1 (Apo A-1), apolipoprotein C-III (Apo C-III), lipid subfractions by nuclear magnetic resonance (NMR) spectroscopy (ie, LDL-C particle size and LDL, very low-density lipoprotein [VLDL], HDL, and intermediate-density lipoprotein [IDL] particle number).
* To assess changes in glycemic parameters with alirocumab vs. usual care treatment.
* To demonstrate the safety and tolerability of alirocumab.
* To evaluate treatment acceptance of alirocumab.
* To evaluate proprotein convertase subtilisin kexin type 9 (PCSK9) concentrations and antibody development.
* To demonstrate the superiority of alirocumab vs. fenofibrate on non-HDL-C and other lipid parameters (subgroup analysis).

DETAILED DESCRIPTION:
The maximum study duration was approximately 9 months per participant, including a 6 month treatment period, a screening period of up to 3 weeks, and an 8 week safety observation period.

For the purpose of scientific communication, a first-step analysis (both efficacy and safety) was performed at the Week 24 cut-off date. A second-step analysis was performed once all participants had completed the study to include a final update of the safety analysis.

ELIGIBILITY:
Inclusion criteria:

* Participants with type 2 diabetes and mixed dyslipidemia whose non-HDL-C was not adequately controlled with a stable, maximum dose/regimen of statin that was tolerated by the participant.
* 18 years of age or more.
* Documented history of atherosclerotic cardiovascular disease (ASCVD) or at least one additional cardiovascular risk factor.
* Non-HDL-C of 100 mg/dL or greater.
* Triglycerides greater than or equal to 150 mg/dL and less than 500 mg/dL.
* Stable anti-hyperglycemic agents for at least 3 months prior to the screening visit and between screening and randomization (including stable insulin dose defined as no variation more than 30% in daily insulin dose within the preceding 3 months, as judged by the Investigator).
* No change in weight of more than 5 kg within the prior 3 months.
* On stable dose of medications that are known to influence weight and/or lipids within the last 3 months.

Exclusion criteria:

* Use of any lipid modifying therapies other than statins within the last 4 weeks (eg, ezetimibe, fenofibrate, nicotinic acid, omega-3 fatty acids, etc.) or use of over the counter products/nutraceuticals known to impact lipids (eg, red yeast rice) within the last 4 weeks.
* Currently drinking more than 2 standard alcoholic drinks per day.
* Body Mass Index (BMI) >45 kg/m² or currently enrolled in a weight loss program and still in active phase of weight loss.
* Glycosylated hemoglobin (HbA1c) 9% or greater.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2016-03-15; Primary Completion 2017-03-22 (Actual); Study Completion 2017-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (119):
- United States (57):
  - Investigational Site Number 840-163, Little Rock, Arkansas
  - Investigational Site Number 840-141, Fresno, California
  - Investigational Site Number 840-152, Huntington Beach, California
  - Investigational Site Number 840-115, La Jolla, California
  - Investigational Site Number 840-118, Los Angeles, California
  - Investigational Site Number 840-106, Northridge, California
  - Investigational Site Number 840-176, Port Hueneme, California
  - Investigational Site Number 840-122, Tarzana, California
  - Investigational Site Number 840-156, Tustin, California
  - Investigational Site Number 840-160, Van Nuys, California
  - Investigational Site Number 840-107, Boca Raton, Florida
  - Investigational Site Number 840-170, Boynton Beach, Florida
  - Investigational Site Number 840-114, Bradenton, Florida
  - Investigational Site Number 840-132, Ocoee, Florida
  - Investigational Site Number 840-179, Oviedo, Florida
  - Investigational Site Number 840-123, Tampa, Florida
  - Investigational Site Number 840-137, Bainbridge, Georgia
  - Investigational Site Number 840-128, Columbus, Georgia
  - Investigational Site Number 840-169, Stockbridge, Georgia
  - Investigational Site Number 840-167, Idaho Falls, Idaho
  - Investigational Site Number 840-161, Chicago, Illinois
  - Investigational Site Number 840-184, Crystal Lake, Illinois
  - Investigational Site Number 840-174, Evanston, Illinois
  - Investigational Site Number 840-138, Springfield, Illinois
  - Investigational Site Number 840-108, Louisville, Kentucky
  - Investigational Site Number 840-183, Paducah, Kentucky
  - Investigational Site Number 840-190, Metairie, Louisiana
  - Investigational Site Number 840-151, Rockville, Maryland
  - Investigational Site Number 840-113, Jefferson City, Missouri
  - Investigational Site Number 840-120, St Louis, Missouri
  - Investigational Site Number 840-148, Omaha, Nebraska
  - Investigational Site Number 840-101, Las Vegas, Nevada
  - Investigational Site Number 840-140, Las Vegas, Nevada
  - Investigational Site Number 840-178, Albany, New York
  - Investigational Site Number 840-181, New York, New York
  - Investigational Site Number 840-157, New York, New York
  - Investigational Site Number 840-188, Greensboro, North Carolina
  - Investigational Site Number 840-131, Morehead City, North Carolina
  - Investigational Site Number 840-158, Morganton, North Carolina
  - Investigational Site Number 840-129, Fargo, North Dakota
  - Investigational Site Number 840-104, Columbus, Ohio
  - Investigational Site Number 840-105, Marion, Ohio
  - Investigational Site Number 840-175, Maumee, Ohio
  - Investigational Site Number 840-136, Bend, Oregon
  - Investigational Site Number 840-187, Murrells Inlet, South Carolina
  - Investigational Site Number 840-111, Summerville, South Carolina
  - Investigational Site Number 840-147, Chattanooga, Tennessee
  - Investigational Site Number 840-159, Knoxville, Tennessee
  - Investigational Site Number 840-153, Dallas, Texas
  - Investigational Site Number 840-143, Houston, Texas
  - Investigational Site Number 840-168, Houston, Texas
  - Investigational Site Number 840-142, Round Rock, Texas
  - Investigational Site Number 840-133, Tomball, Texas
  - Investigational Site Number 840-185, Orem, Utah
  - Investigational Site Number 840-150, Salt Lake City, Utah
  - Investigational Site Number 840-126, Chesapeake, Virginia
  - Investigational Site Number 840-171, Richmond, Virginia
- Australia (3):
  - Investigational Site Number 036102, Herston
  - Investigational Site Number 036104, Merewether
  - Investigational Site Number 036101, St Leonards
- Brazil (6):
  - Investigational Site Number 076103, Campinas
  - Investigational Site Number 076104, Fortaleza
  - Investigational Site Number 076105, São Paulo
  - Investigational Site Number 076101, São Paulo
  - Investigational Site Number 076106, São Paulo
  - Investigational Site Number 076102, São Paulo
- Finland (3):
  - Investigational Site Number 246102, Oulu
  - Investigational Site Number 246101, Oulu
  - Investigational Site Number 246104, Tampere
- Germany (10):
  - Investigational Site Number 276112, Berlin
  - Investigational Site Number 276109, Berlin
  - Investigational Site Number 276104, Dippoldiswalde
  - Investigational Site Number 276101, Dresden
  - Investigational Site Number 276110, Essen
  - Investigational Site Number 276108, Essen
  - Investigational Site Number 276111, Goch
  - Investigational Site Number 276107, Karlsruhe
  - Investigational Site Number 276103, Künzing
  - Investigational Site Number 276102, Oldenburg in Holstein
- Israel (5):
  - Investigational Site Number 376101, Beersheba
  - Investigational Site Number 376103, Petah Tikva
  - Investigational Site Number 376104, Petah Tikva
  - Investigational Site Number 376102, Rehovot
  - Investigational Site Number 376106, Tel Aviv
- Italy (8):
  - Investigational Site Number 380104, Bergamo
  - Investigational Site Number 380107, Catanzaro
  - Investigational Site Number 380103, Napoli
  - Investigational Site Number 380108, Padua
  - Investigational Site Number 380106, Partinico
  - Investigational Site Number 380101, Pisa
  - Investigational Site Number 380105, Roma
  - Investigational Site Number 380102, Torino
- Investigational Site Number 414101, Kuwait City, Kuwait
- Lebanon (2):
  - Investigational Site Number 422101, Beirut
  - Investigational Site Number 422102, Hazmiyeh
- Norway (2):
  - Investigational Site Number 578101, Oslo
  - Investigational Site Number 578102, Oslo
- Sweden (2):
  - Investigational Site Number 752102, Gothenburg
  - Investigational Site Number 752101, Stockholm
- Switzerland (3):
  - Investigational Site Number 756101, Geneva
  - Investigational Site Number 756102, Olten
  - Investigational Site Number 756103, Reinach
- Turkey (Türkiye) (10):
  - Investigational Site Number 792105, Adana
  - Investigational Site Number 792106, Ankara
  - Investigational Site Number 792102, Ankara
  - Investigational Site Number 792108, Çorum
  - Investigational Site Number 792109, Hatay
  - Investigational Site Number 792104, Izmir
  - Investigational Site Number 792101, Izmir
  - Investigational Site Number 792110, Izmir
  - Investigational Site Number 792107, Kayseri
  - Investigational Site Number 792103, Samsun
- Investigational Site Number 784101, Dubai, United Arab Emirates
- United Kingdom (6):
  - Investigational Site Number 826104, Exeter
  - Investigational Site Number 826106, Manchester
  - Investigational Site Number 826105, Middlesbrough
  - Investigational Site Number 826103, Stevenage
  - Investigational Site Number 826101, Torquay
  - Investigational Site Number 826102, West Bromwich

REFERENCES:
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- [Derived] Colhoun HM, Leiter LA, Muller-Wieland D, Cariou B, Ray KK, Tinahones FJ, Domenger C, Letierce A, Israel M, Samuel R, Del Prato S. Effect of alirocumab on individuals with type 2 diabetes, high triglycerides, and low high-density lipoprotein cholesterol. Cardiovasc Diabetol. 2020 Feb 8;19(1):14. doi: 10.1186/s12933-020-0991-1. PMID 32035487
- [Derived] Ray KK, Del Prato S, Muller-Wieland D, Cariou B, Colhoun HM, Tinahones FJ, Domenger C, Letierce A, Mandel J, Samuel R, Bujas-Bobanovic M, Leiter LA. Alirocumab therapy in individuals with type 2 diabetes mellitus and atherosclerotic cardiovascular disease: analysis of the ODYSSEY DM-DYSLIPIDEMIA and DM-INSULIN studies. Cardiovasc Diabetol. 2019 Nov 9;18(1):149. doi: 10.1186/s12933-019-0951-9. PMID 31706300
- [Derived] Ray KK, Leiter LA, Muller-Wieland D, Cariou B, Colhoun HM, Henry RR, Tinahones FJ, Bujas-Bobanovic M, Domenger C, Letierce A, Samuel R, Del Prato S. Alirocumab vs usual lipid-lowering care as add-on to statin therapy in individuals with type 2 diabetes and mixed dyslipidaemia: The ODYSSEY DM-DYSLIPIDEMIA randomized trial. Diabetes Obes Metab. 2018 Jun;20(6):1479-1489. doi: 10.1111/dom.13257. Epub 2018 Mar 23. PMID 29436756
- [Derived] Muller-Wieland D, Leiter LA, Cariou B, Letierce A, Colhoun HM, Del Prato S, Henry RR, Tinahones FJ, Aurand L, Maroni J, Ray KK, Bujas-Bobanovic M. Design and rationale of the ODYSSEY DM-DYSLIPIDEMIA trial: lipid-lowering efficacy and safety of alirocumab in individuals with type 2 diabetes and mixed dyslipidaemia at high cardiovascular risk. Cardiovasc Diabetol. 2017 May 25;16(1):70. doi: 10.1186/s12933-017-0552-4. PMID 28545518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 119 centers in 15 countries. A total of 864 participants were screened between March 2016 and September 2016, 451 of whom were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: Randomization was stratified by investigator's choice of usual care therapy, which was pre-specified prior to randomization. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 2:1 ratio (alirocumab: usual care) after confirmation of selection criteria. 413 participants were randomized.
Groups:
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: Alirocumab 75 mg subcutaneous (SC) injection every 2 weeks (Q2W) added to insulin or other antihyperglycemic drugs, stable maximally tolerated dose of statin therapy without other lipid modifying therapies (LMT) for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when non-high-density lipoprotein cholesterol (non-HDL-C) levels >=100 mg/dL (2.59 mmol/L) at Week 8.
Period: Overall Study
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Started | 276 (Randomized) | 137 (Randomized)
Treated (Safety Population) | 275 | 137
ITT Population | 273 | 136
ITT: Intent to Prescribe Fenofibrate | 47 (Fenofibrate was only 'intended to prescribe' in the Alirocumab arm but not actually administered.) | 24
Completed (Completed = treatment completion) | 245 | 129
Not Completed | 31 | 8
Not completed — Randomized but not treated | 1 | 0
Not completed — Adverse Event | 10 | 4
Not completed — Withdrawal by Subject | 9 | 1
Not completed — Poor compliance to study protocol | 1 | 0
Not completed — Other than specified above | 10 | 3

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Alirocumab 75 mg Q2W/Up to 150 mg Q2W: Alirocumab 75 mg SC injection Q2W added to insulin or other antihyperglycemic drugs, stable maximally tolerated dose of statin therapy without other LMT for 24 weeks. Alirocumab dose up-titrated to 150 mg Q2W from Week 12 when non-HDL-C levels >=100 mg/dL (2.59 mmol/L) at Week 8.
- Total: Total of all reporting groups
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care | Total
Number analyzed (Participants) | 276 | 137 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.3) | 64.1 (8.8) | 63.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 68 | 197
  Male | 147 | 69 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 14 | 49
  Not Hispanic or Latino | 240 | 123 | 363
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 247 | 123 | 370
  Black | 16 | 6 | 22
  Asian/Oriental | 3 | 7 | 10
  American Indian or Alaska Native | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 6 | 1 | 7
Non-HDL-C [Mean (Standard Deviation); unit: mg/dL] — non-HDL-C = Total cholesterol (Total-C) minus high-density lipoprotein cholesterol (HDL-C)
  mg/dL | 155.1 (46.2) | 161.5 (48.8) | 157.2 (47.1)
Non-HDL-C [Mean (Standard Deviation); unit: mmol/L] — non-HDL-C = Total-C minus HDL-C
  mmol/L | 4.0 (1.2) | 4.2 (1.2) | 4.073 (1.221)
Intent to Prescribe Treatment [Count of Participants; unit: Participants] — Randomization was stratified by the Investigator's selection of usual care therapy prior to randomization. LMTs were only 'intended to prescribe' in the Alirocumab arm but not actually administered.
  Participants
    Fenofibrate | 48 | 24 | 72
    No additional LMT | 79 | 39 | 118
    Ezetimibe | 104 | 52 | 156
    Omega-3 fatty acids | 43 | 21 | 64
    Nicotinic acid | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24: Overall Intent-to-treat (ITT) Analysis
Description: Adjusted Least-squares (LS) means and standard errors at Week 24 were obtained from a mixed-effect model with repeated measures (MMRM) to account for missing data. All available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment were used in the model (ITT analysis).
Time Frame: From Baseline to Week 24
Population: ITT population: all randomized participants with one baseline and at least one post-baseline non-HDL-C value on- or off-treatment.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | -37.3 (3.0) | -4.7 (3.3)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care; Alirocumab group was compared to usual care group using an appropriate contrast statement; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -32.5, 97.5% CI 2-sided [-38.1 to -27.0] — Alirocumab vs. usual care

2. Primary Outcome: Percent Change From Baseline in Non-HDL-C at Week 24: ITT- Intent to Prescribe Fenofibrate Stratum
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment in the intent to prescribe fenofibrate stratum. The usual care here corresponds to fenofibrate.
Time Frame: From Baseline to Week 24
Population: ITT population. Here, 'Number of participants analyzed' = participants from intent to prescribe fenofibrate stratum who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Usual Care: Intent to Prescribe Fenofibrate: Participants on usual care continued on insulin or other antihyperglycemic drugs, stable maximally tolerated dose of statin therapy with fenofibrate as per Investigator's judgment for 24 weeks.
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | -41.7 (3.4) | -8.5 (4.8)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care: Intent to Prescribe Fenofibrate; Alirocumab group was compared to usual care group for the intent to prescribe fenofibrate using an appropriate contrast statement; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -33.3, 97.5% CI 2-sided [-46.6 to -19.9] — Alirocumab (intent to prescribe fenofibrate) vs. usual care (intent to prescribe fenofibrate)

3. Secondary Outcome: Percent Change From Baseline in Measured Low-Density Lipoprotein Cholesterol (LDL-C) at Week 24: Overall ITT Analysis
Description: Measured LDL-C values via beta quantification method. Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline LDL-C value on-or off-treatment (LDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | -43.3 (3.6) | -0.3 (4.0)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses for overall ITT analysis. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -43.0, 97.5% CI 2-sided [-49.7 to -36.3] — Alirocumab vs. usual care

4. Secondary Outcome: Percent Change From Baseline in Measured LDL-C at Week 24: ITT- Intent to Prescribe Fenofibrate Stratum
Description: Measured LDL-C values via beta quantification method. Adjusted LS means and standard errors at Week 24 from MMRM model including available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment in the intent to prescribe fenofibrate stratum. The usual care here corresponds to fenofibrate.
Time Frame: From Baseline to Week 24
Population: LDL-C ITT population. Here, 'Number of participants analyzed' = participants from intent to prescribe fenofibrate stratum who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | -47.0 (4.2) | 8.7 (5.8)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care: Intent to Prescribe Fenofibrate; A separate hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses for ITT-intent to prescribe fenofibrate stratum. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -55.7, 97.5% CI 2-sided [-71.8 to -39.6] — Alirocumab (intent to prescribe fenofibrate) vs. usual care (intent to prescribe fenofibrate)

5. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12: Overall ITT Analysis
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | -35.5 (2.9) | -9.4 (3.2)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care; Testing according to the hierarchical testing procedure (only performed if the previous endpoint of overall ITT analysis was statistically significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -26.1, 97.5% CI 2-sided [-31.5 to -20.7] — Alirocumab vs. usual care

6. Secondary Outcome: Percent Change From Baseline in Non-HDL-C at Week 12: ITT- Intent to Prescribe Fenofibrate Stratum
Description: Adjusted LS means and standard errors at Week 12 from MMRM model including all available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment in the intent to prescribe fenofibrate stratum. The usual care here corresponds to fenofibrate.
Time Frame: From Baseline to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | -34.7 (3.2) | -7.3 (4.5)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care: Intent to Prescribe Fenofibrate; Testing according to the hierarchical testing procedure (only performed if the previous endpoint of ITT-intent to prescribe fenofibrate stratum was statistically significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -27.4, 97.5% CI 2-sided [-40.0 to -14.8] — Alirocumab (intent to prescribe fenofibrate) vs. usual care (intent to prescribe fenofibrate)

7. Secondary Outcome: Percent Change From Baseline in Measured LDL-C at Week 12: Overall ITT Analysis
Description: Measured LDL-C values via beta quantification method. Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: LDL-C ITT population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | -41.7 (3.3) | -7.0 (3.6)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -34.7, 97.5% CI 2-sided [-40.8 to -28.6] — Alirocumab vs. usual care

8. Secondary Outcome: Percent Change From Baseline in Measured LDL-C at Week 12: ITT- Intent to Prescribe Fenofibrate Stratum
Description: Measured LDL-C values via beta quantification method. Adjusted LS means and standard errors at Week 12 from MMRM model including available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment in the intent to prescribe fenofibrate stratum. The usual care here corresponds to fenofibrate.
Time Frame: From Baseline to Week 24
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | -44.3 (3.6) | 5.4 (5.1)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care: Intent to Prescribe Fenofibrate; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -49.7, 97.5% CI 2-sided [-63.7 to -35.8] — Alirocumab (intent to prescribe fenofibrate) vs. usual care (intent to prescribe fenofibrate)

9. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo-B) at Week 24: Overall ITT Analysis
Description: Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Apo-B value on-or off-treatment (Apo-B ITT population).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | -33.8 (2.7) | -1.6 (3.0)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -32.3, 97.5% CI 2-sided [-37.3 to -27.2] — Alirocumab vs. usual care

10. Secondary Outcome: Percent Change From Baseline in Apo B at Week 24: ITT- Intent to Prescribe Fenofibrate Stratum
Description: as for outcome 2
Time Frame: From Baseline to Week 24
Population: Apo-B ITT population.Here, 'Number of participants analyzed' = participants from intent to prescribe fenofibrate stratum who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | -38.9 (3.1) | -3.8 (4.4)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care: Intent to Prescribe Fenofibrate; Testing according to the hierarchical testing procedure (only performed if the previous endpoint of ITT- intent to prescribe fenofibrate stratum was statistically significant); Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -35.2, 97.5% CI 2-sided [-47.4 to -22.9] — Alirocumab (intent to prescribe fenofibrate) vs. usual care (intent to prescribe fenofibrate)

11. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Total-C) at Week 24 : Overall ITT Analysis
Description: as for outcome 9
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline Total-C value on- or off-treatment (Total-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | -27.4 (2.3) | -2.8 (2.5)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -24.6, 97.5% CI 2-sided [-28.8 to -20.3] — Alirocumab vs. usual care

12. Secondary Outcome: Percent Change From Baseline in Total-C at Week 24: ITT- Intent to Prescribe Fenofibrate Stratum
Description: as for outcome 2
Time Frame: From Baseline to Week 24
Population: Total-C ITT population. Here, 'Number of participants analyzed' = participants from intent to prescribe fenofibrate stratum who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | -30.9 (2.6) | -5.7 (3.7)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care: Intent to Prescribe Fenofibrate; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Threshold for significance <=0.025; LS Mean Difference = -25.3, 97.5% CI 2-sided [-35.4 to -15.1] — Alirocumab (intent to prescribe fenofibrate) vs. usual care (intent to prescribe fenofibrate)

13. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24 : Overall ITT Analysis
Description: Adjusted means and standard errors at Week 24 were obtained from multiple imputation approach followed by robust regression model for handling of missing data. All available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment were included in the imputation model.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | -23.7 (1.9) | 3.7 (2.6)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Regression, Robust — Threshold for significance <=0.025; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -27.4, 97.5% CI 2-sided [-34.6 to -20.1] — Alirocumab vs. usual care

14. Secondary Outcome: Percent Change From Baseline in Lipoprotein(a) at Week 24: ITT- Intent to Prescribe Fenofibrate Stratum
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment in the intent to prescribe fenofibrate stratum. The usual care here corresponds to fenofibrate.
Time Frame: From Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | -18.9 (4.4) | 3.9 (6.6)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care: Intent to Prescribe Fenofibrate; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.0040, Regression, Robust — Threshold for significance <=0.025; Multiple imputation approach followed by robust regression model; Adjusted Mean Difference = -22.8, 97.5% CI 2-sided [-40.6 to -5.0] — Alirocumab (intent to prescribe fenofibrate) vs. usual care (intent to prescribe fenofibrate)

15. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24: Overall ITT Analysis
Description: Adjusted means and standard errors at Week 24 from multiple imputation approach followed by robust regression model including all available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: ITT population.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | -13.0 (2.0) | -8.8 (2.8)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.2191, Regression, Robust — Threshold for significance <=0.025; Multiple imputation approach followed by robust regression; Adjusted Mean Difference = -4.2, 97.5% CI 2-sided [-11.8 to 3.4] — Alirocumab vs. usual care

16. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides at Week 24: ITT- Intent to Prescribe Fenofibrate Stratum
Description: as for outcome 14
Time Frame: From Baseline to Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | -15.4 (4.7) | -24.4 (6.6)
Statistical Analysis 1: Comparison: Alirocumab 75 mg Q2W/Up to 150 mg Q2W vs Usual Care: Intent to Prescribe Fenofibrate; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.2651, Regression, Robust — Threshold for significance <=0.025; Multiple imputation approach followed by robust regression; Adjusted Mean Difference = 9.0, 97.5% CI 2-sided [-9.1 to 27.1]; Alirocumab (intent to prescribe fenofibrate) vs. usual care (intent to prescribe fenofibrate)

17. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24 : Overall ITT Analysis
Description: as for outcome 9
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline HDL-C value on- or off-treatment (HDL-C ITT population).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Percent change | 14.5 (2.5) | 8.2 (2.7)

18. Secondary Outcome: Percent Change From Baseline in HDL-C at Week 24: ITT- Intent to Prescribe Fenofibrate Stratum
Description: as for outcome 2
Time Frame: From Baseline to Week 24
Population: HDL-C ITT population. Here, 'Number of participants analyzed' = participants from intent to prescribe fenofibrate stratum who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 47 | 24
Percent change | 13.5 (2.9) | 12.3 (4.1)

19. Secondary Outcome: Percent Change From Baseline in LDL-C Particle Number at Week 24: Overall ITT Analysis
Description: LDL-C particle number was calculated from lipid subfractions by nuclear magnetic resonance (NMR) spectroscopy. Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment.
Time Frame: From Baseline to Week 24
Population: Participants of the ITT population with one baseline and at least one post-baseline LDL-C particle number on- or off-treatment (LDL-C particle number ITT population).
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 270 | 135
Percent change | -41.6 (3.0) | -3.9 (3.4)

20. Secondary Outcome: Percent Change From Baseline in LDL-C Particle Number at Week 24: ITT- Intent to Prescribe Fenofibrate Stratum
Description: LDL-C particle number was calculated from lipid subfractions by NMR spectroscopy. Adjusted LS means and standard errors at Week 24 from MMRM model including all available post-baseline data from Week 8 to Week 24 regardless of status on- or off-treatment in the intent to prescribe fenofibrate stratum. The usual care here corresponds to fenofibrate.
Time Frame: From Baseline to Week 24
Population: LDL-C particle number ITT population. Here, 'Number of participants analyzed' = participants from intent to prescribe fenofibrate stratum who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care: Intent to Prescribe Fenofibrate
Number analyzed (Participants) | 46 | 24
Percent change | -45.4 (3.5) | -2.9 (5.0)

21. Secondary Outcome: Absolute Change From Baseline in Hemoglobin A1c (HbA1c) at Week 12 and 24 : Overall ITT Analysis
Description: Absolute change = HbA1c value at specified week minus HbA1c value at baseline.
Time Frame: Baseline, Week 12 and 24
Population: ITT population. Here, 'Number Analyzed' = participants with available data at the specified time points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
mmol/mol
  Change at Week 12: number analyzed (Participants) | 265 | 133
  Change at Week 12 | 0.59 (6.82) | 0.43 (5.70)
  Change at Week 24: number analyzed (Participants) | 251 | 128
  Change at Week 24 | 2.84 (8.04) | 2.40 (8.19)

22. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) at Week 12 and 24 : Overall ITT Analysis
Description: Absolute change = FPG value at specified week minus FPG value at baseline.
Time Frame: Baseline, Week 12 and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
mmol/L
  Change at Week 12: number analyzed (Participants) | 262 | 133
  Change at Week 12 | 0.45 (2.43) | 0.21 (1.86)
  Change at Week 24: number analyzed (Participants) | 251 | 128
  Change at Week 24 | 0.68 (2.54) | 0.03 (2.54)

23. Secondary Outcome: Absolute Change From Baseline in Number of Glucose-Lowering Treatments at Week 12 and 24 : Overall ITT Analysis
Description: Glucose lowering treatment was calculated for non-insulin treatments as one for each unique treatment received and for insulin treatment as one in total for all participants who have taken one or more treatments. Absolute change = number of glucose-lowering treatments at specified week minus baseline value.
Time Frame: Baseline, Week 12 and 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Glucose lowering treatments
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
Number analyzed (Participants) | 273 | 136
Glucose lowering treatments
  Change at Week 12: number analyzed (Participants) | 271 | 136
  Change at Week 12 | 0.04 (0.30) | 0.04 (0.19)
  Change at Week 24: number analyzed (Participants) | 267 | 135
  Change at Week 24 | 0.07 (0.37) | 0.04 (0.23)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 32) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are TEAEs that are AEs that developed/worsened and death that occurred during the 'treatment-emergent period' (the time from the first dose of study drug up to the last dose of study drug +70 days).
Arm/Group | Alirocumab 75 mg Q2W/Up to 150 mg Q2W | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/275 | 0/137
Serious Adverse Events (participants affected / at risk) | 26/275 | 12/137
Other Adverse Events (participants affected / at risk) | 37/275 | 27/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (N=275) | Usual Care (N=137)
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 3 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 2
Seizure (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alirocumab 75 mg Q2W/Up to 150 mg Q2W (N=275) | Usual Care (N=137)
Diarrhoea (Gastrointestinal disorders) | 14 | 9
Bronchitis (Infections and infestations) | 5 | 7
Urinary tract infection (Infections and infestations) | 15 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/59/NCT02642159/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT02642159/SAP_001.pdf